CLINICAL TRIAL: NCT03391180
Title: The Effect of ICON Treatment on WPL With Patients After Fixed Orthodontic Appliances: A Randomized Controlled Trial
Brief Title: The Effect of ICON Treatment on WPL With Patients After Fixed Orthodontic Appliances
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Riyadh Colleges of Dentistry and Pharmacy (Other)
Responsible Party: Principal Investigator, Omar Alkadhi, Lecturer, Riyadh Colleges of Dentistry and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FGR/2018/45
Record Dates: First submitted 2017-12-26; First posted 2018-01-05 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: White Spot Lesion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICON Remineralization (Experimental): Firstly, Conditioning of the WSL surface by 15% HCL gel (Icon-Etch, DNG) and subsequent application of the drying solution (Icon-Dry, DMG), Numbers of additional etching intervals have been determined by visual assessment after each of the etch/dry intervals to achieve individual, customized intensities of WSL surface conditioning.
  Interventions: Drug: ICON Remineralization
- CPP-ACPF (Active Comparator): Participants in group 2 (CPP-ACPF) were treated with applying a pea sized amount of ACC-ACPF plus on a gloved finger of the examiner and rubbed the surface of the labial tooth for 4 minutes with advising the patient to avoid drinking and eating for the next 30 minutes of application.
  Interventions: Drug: CPP-ACPF

INTERVENTIONS:
Drug: ICON Remineralization — A material used for the Remineralization of white spot lesions.
  Arms: ICON Remineralization
Drug: CPP-ACPF — Casein phosphopeptide-Amorphous calcium phosphate fluoride used for the remineralization of white spot lesions.
  Arms: CPP-ACPF

SUMMARY:
The aim of this study is to determine the effect of ICON on White spot lesions compared to CPP-ACPF plus.

DETAILED DESCRIPTION:
The participants were categorized to either group (group1) receiving ICON treatment method (Icon, DMG, Germany), or (group 2) who shall be receiving CPP-ACPF treatment method (Tooth Mousse plus).

ELIGIBILITY:
Inclusion Criteria:

* permanent dentition, in good general health and without systemic diseases, who had received fixed orthodontic treatment.

Exclusion Criteria:

* Patients with primary dentition, enamel hypoplasia, dental fluorosis or tetracycline pigmentation and carious cavity were excluded.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-02 (Estimated); Primary Completion 2018-04 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Remineralization | 3 Months
  Using DIAGNOdent Laser device.

CONTACTS AND LOCATIONS:
Overall Officials: Omar H AlKadhi, Principal Investigator — Riyadh Colleges of Dentistry and Pharmacy
Locations (1):
- Riyadh Colleges of Dentistry and Pharmacy, Riyadh, ArRiyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No